CLINICAL TRIAL: NCT01991561
Title: Immunogenicity, Safety, Tolerability of a Plant-made H5 VLP Influenza Vaccine.
Brief Title: Immunogenicity, Safety, Tolerability of a Plant-made H5 Virus-like-particle (VLP) Influenza Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicago (Industry)
Collaborators: Syneos Health (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-H5VLP-005
Record Dates: First submitted 2013-09-18; First posted 2013-11-25 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2015-09

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Influenza, Human; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Aluminum Hydroxide; Adjuvants, Immunologic; Immunogenic Factors; GLA-SE; Physiological Effects of Drugs; Virus Diseases; Orthomyxoviridae Infections; Infection
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections; Infections | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Low dose of H5 VLP vaccine + Alhydrogel (Experimental): Biological: low dose of H5 VLP vaccine 2 doses given 21 days apart of low dose of H5 VLP vaccine mixed with Alhydrogel
  Interventions: Biological: Low dose of H5 VLP vaccine + Alhydrogel
- Med dose H5 VLP vaccine + Alhydrogel (Experimental): Biological:Med dose of H5 VLP vaccine + Alhydrogel, 2 doses given 21 days apart of Med dose H5 VLP vaccine mixed with Alhydrogel
  Interventions: Biological: Med dose of H5 VLP vaccine + Alhydrogel
- High dose of H5 VLP vaccine + Alhydrogel (Experimental): Biological: High dose of H5 VLP vaccine 2 doses given 21 days apart of High dose of H5 VLP vaccine mixed with Alhydrogel
  Interventions: Biological: High dose of H5 VLP vaccine + Alhydrogel
- Low dose of H5 VLP vaccine + GLA-SE (Experimental): Biological: low dose of H5 VLP vaccine 2 doses given 21 days apart of low dose of H5 VLP vaccine mixed with GLA-SE
  Interventions: Biological: Low dose of H5 VLP vaccine + GLA-SE
- High dose of H5 VLP vaccine + GLA-SE (Experimental): Biological: High dose of H5 VLP vaccine 2 doses given 21 days apart of High dose of H5 VLP vaccine mixed with GLA-SE
  Interventions: Biological: High dose of H5 VLP vaccine + GLA-SE
- Placebo comparator: Placebo (Placebo Comparator): Biological: Placebo 2 doses given 21 days apart of the placebo
  Interventions: Biological: Placebo comparator: Placebo

INTERVENTIONS:
Biological: Low dose of H5 VLP vaccine + Alhydrogel — Biological: low dose of H5 VLP vaccine 2 doses given 21 days apart of low dose of H5 VLP vaccine mixed with Alhydrogel
  Arms: Low dose of H5 VLP vaccine + Alhydrogel
Biological: Med dose of H5 VLP vaccine + Alhydrogel — Biological:Med dose of H5 VLP vaccine 2 doses given 21 days apart of Med dose H5 VLP vaccine mixed with Alhydrogel
  Arms: Med dose H5 VLP vaccine + Alhydrogel
Biological: High dose of H5 VLP vaccine + Alhydrogel — Biological: High dose of H5 VLP vaccine 2 doses given 21 days apart of High dose of H5 VLP vaccine mixed with Alhydrogel
  Arms: High dose of H5 VLP vaccine + Alhydrogel
Biological: Low dose of H5 VLP vaccine + GLA-SE — Biological: low dose of H5 VLP vaccine 2 doses given 21 days apart of low dose of H5 VLP vaccine mixed with GLA-SE
  Arms: Low dose of H5 VLP vaccine + GLA-SE
Biological: High dose of H5 VLP vaccine + GLA-SE — Biological: High dose of H5 VLP vaccine 2 doses given 21 days apart of High dose of H5 VLP vaccine mixed with GLA-SE
  Arms: High dose of H5 VLP vaccine + GLA-SE
Biological: Placebo comparator: Placebo — Biological: Placebo 2 doses given 21 days apart of the placebo
  Arms: Placebo comparator: Placebo

SUMMARY:
A phase 2, Randomized, Observer-blind, Multicenter, Dose-Ranging Study to Evaluate the Immunogenicity, Safety, and Tolerability of the plant-made H5 VLP Influenza vaccine adjuvanted with Alhydrogel or Glucopyranosyl-lipid adjuvant in squalene emulsion (GLA-SE), in healthy adults 18-60 years of age.

DETAILED DESCRIPTION:
This study will consist of a dose-ranging in 390 subjects who will be randomized to receive one injection at Days 0 and 21 of either a low, medium or a high dose of H5 VLP Influenza vaccine combined with Alhydrogel®, or a low or high dose of H5 VLP Influenza vaccine combined with GLA-SE, or the placebo preparation (100 millimolar (mM) phosphate buffer + 150 mM Sodium Chloride (NaCl) + 0.01% Tween 80). Seven-day (7) safety data after the first immunization of the first 25% study subjects enrolled (98 subjects) will be tabulated and reviewed by the Data and Safety Monitoring Board (DSMB), prior to permitting the first immunization of the remaining study subjects and the second immunisations. Also, based on medical expert opinion and on safety criteria defined in the protocol, a DSMB review might be necessary on the seven-day safety data of the same 25% study subjects following administration of their second dose, before proceeding to the second immunizations of the remaining study subjects. Twenty-one (21) days after each immunization, key safety and immunogenicity data will be collected and analysed. All subjects will be followed for safety until Day 407.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults, 18 to 60 years of age, inclusive
2. Healthy as judged by the Investigator and determined by medical history, history/symptom-directed physical examination, vital signs, screening laboratories and medical history conducted no more than 30 days prior to study vaccine administration;
3. BMI of ≥18 and ≤ 32;
4. Comprehension of the study requirements, expressed availability for the required study period and ability to attend scheduled visits;
5. Accessible by telephone on a regular basis;
6. In the opinion of the Investigator, ability and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee;
7. If female, have a negative serum pregnancy test result at study entry, and if capable of child bearing has been consistently using effective birth control for the 28 days prior to study entry and agree to continue employing adequate birth control measures for the duration of the study.

Exclusion Criteria:

1. Presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

   1. Requiring a new medical or surgical treatment within one month prior to study vaccine administration;
   2. Requiring a change in medication dosage in one month prior to test article administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
   3. Hospitalization or an event fulfilling the definition of a serious adverse event within one month prior to test article administration;
2. Any medical or neuropsychiatric condition which, in the Investigator's opinion, would render the subject unable to provide informed consent or unable to provide valid safety observations and reporting;
3. Any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection or Hepatitis B or C or presence of lymphoproliferative disease;
4. Presence of any febrile illness, oral temperature of >38.0˚C within 24 hours of test article administration. Such subjects may be re-evaluated for enrolment after resolution of illness;
5. History of autoimmune disease;
6. Administration of any vaccine (including any other influenza vaccine) within a 30 day period prior to study enrolment, or planned administration within the period from the first vaccination up to blood sampling at Day 42 or within 30 days prior to blood sampling at Day 228. Immunization on an emergency basis of a tetanus and diphtheria toxoids adsorbed for adult use (Td) will be allowed provided the vaccine is not administered within two weeks prior to test article administration. Receipt of any other emergency immunizations (e.g. rabies) will result in a case-by-case review of continued participation;
7. Use of any investigational or non-registered product within 30 days prior to study enrolment or planned use during the study period. Subjects may not participate in any other drug study while participating in this study;
8. Treatment with systemic glucocorticoids at a dose exceeding ≥ 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of first test article administration, or any other cytotoxic or immunosuppressant drug or any immune globulin preparation within three months of vaccination. Nasal or inhaled glucocorticoids are allowed;
9. Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin, and without a clinically apparent bleeding tendency are eligible;
10. History of previous H5N1 vaccination or a history of exposure to H5N1 virus. Any subject that was enrolled on our previous H5 studies (except the ones that received placebo) would not be eligible;
11. Are at high risk of contracting H5N1 influenza infection (e.g. poultry workers);
12. History of allergy to any of the constituents of H5 VLP (H5N1) study vaccine, Alhydrogel® (aluminum hydroxide), GLA-SE, or the phosphate buffer;
13. History of severe allergic reactions (including anaphylaxis) to any food, medication, or bee sting or previous status of asthmatic;
14. History of tobacco allergy;
15. History of egg allergy (). GLA-SE contains egg phosphatidylcholine.
16. Continuous use of anti-histamines in last 4 weeks prior to immunization and use of antihistamine in last 48 hours prior to immunization;
17. Have a rash, dermatological condition or tattoos or a muscle mass condition at the injection site that may interfere with injection site reaction rating. ;
18. Have received a blood transfusion or immunoglobulins within 90 days of study entry;
19. If female, and of childbearing potential, has not been consistently using effective birth control for the 28 days prior to study entry. An example of highly effective birth control is oral contraceptives, hormone implants, abstinence (self-reported), or male condom plus spermicide. All female subjects, regardless of birth control history must provide a serum sample for pregnancy screening. Effective birth control must be used for the duration of the study for female of child bearing potential. The subject must have no plan to become pregnant during the study period;
20. Among female subjects, either known pregnancy or urine beta-human chorionic gonadotropin (ß-hCG) test results consistent with pregnancy prior to test article administration on Day 0 and 21;
21. Female subjects who are lactating;
22. Vital sign abnormalities: systolic blood pressure >150 mmHg, diastolic blood pressure >90 mmHg, resting pulse rate <40 bpm or >100 bpm or according to the Investigator's opinion;
23. Cancer or treatment for cancer within 3 years of test article administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Levels of antibodies induced against the H5 of the H5N1/A/Indonesia/5/05, clade 2.1 virus | 21 days after each injection
  Immunogenicity Geometric mean titers (GMTs) of hemagglutination inhibition (HI antibody on Day 21).
Levels of antibodies induced against the H5 of the H5N1/A/Indonesia/5/05, clade 2.1 virus | 42 days after each injection
  Immunogenicity Geometric mean titers (GMTs) of hemagglutination inhibition (HI antibody on Day 42).

SECONDARY OUTCOMES:
Cross-reactivity of antibodies induced by 2 consecutive doses of H5 VLP influenza vaccine | 21 days after each injection
  Measures of Geometric Mean Fold Rise, seroconversion rate and seroprotection rate (for HI only).
Reactivity of antibodies induced by 2 consecutive doses of H5 VLP influenza vaccine given 21 days apart | 21 days after each injection
  GMFR, seroconversion rate, percentage of subjects with a detectable MN antibody response

CONTACTS AND LOCATIONS:
Overall Officials: Michael Libman, MD, Principal Investigator — MUHC-Vaccine Study Centre; Luis Robles, MD, Principal Investigator — Syneos Health
Locations (2):
- Canada (2):
  - INC Research, Toronto, Ontario
  - MUHC Vaccine Study Center, Pierrefonds, Quebec